CLINICAL TRIAL: NCT03739346
Title: Efficacy of Hypnosis Compared With Tell/Show/do Technique in Anxiety/Pain Reduction in Children During Pulpotomies
Brief Title: Efficacy of Hypnosis in Anxiety/Pain Reduction in Children During Pulpotomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alejandra Ramírez Carrasco (Other)
Responsible Party: Sponsor-Investigator, Alejandra Ramírez Carrasco, Principal Investigator, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIFE-032-017
Record Dates: First submitted 2018-09-11; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Dental Anxiety; Pain
Keywords: Dental anxiety; Pain; Child; Pediatric dentistry; Hypnosis
MeSH Terms: conditions — Pain | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Tell, show, do technique
  Interventions: Behavioral: Tell, show, do technique
- Intervention (Experimental): Hypnosis.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — Therapeutic technique in which clinicians make suggestions to individuals who have undergone a procedure designed to relax them and focus their minds.
  Arms: Intervention
Behavioral: Tell, show, do technique — The technique involves verbal explanations of procedures in phrases appropriate to the developmental level of the patient (tell); demonstrations for the patient of the visual, auditory, olfactory, and tactile aspects of the procedure in a carefully defined, nonthreatening setting (show); and then, without deviating from the explanation and demonstration, completion of the procedure (do). Tell-show-do technique is used with communication skills (verbal and nonverbal) and positive reinforcement.
  Arms: Control

SUMMARY:
Anxiety and pain are emotions that the child often experiences in the dental office, generating the appearance of negative, uncooperative and even disruptive behaviors during the treatment; these make it difficult for dental care and the possibility of establishing a relationship of trust between the pediatric dentist and the patient. The pediatric dentist must promote a positive attitude of the child throughout the dental treatment, keep the child calm and avoid feeling pain is essential at each appointment.

When carrying out dental treatments that are more invasive or painful for the patient, such as pulpotomies, it is difficult to distinguish and separate anxiety from pain.

In this project, anxiety/pain will be managed as a whole, to assess it with the same scale, and to correlate the scores obtained with the variations in skin conductance and heart rate, before, during and after perform pulpotomies in children.

ELIGIBILITY:
Inclusion Criteria:

* Without previous dental experiences, patients with clinical and radiographic indication of pulpotomy in at least one temporary inferior molar, clinically healthy patients, patients whose parents accept entry into the study and who sign the informed consent.

Exclusion Criteria:

* Patients who have received hypnosis before.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability Scale | Change from score in baseline at score during pulpotomies and after pulpotomies, through study completation average 3 months.
  A measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
  Each category is scored on the 0-2 scale which results in a total score of 0-10. 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Pierdant Pérez, Master, Study Director — Universidad Autonoma de San Luis Potosí

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appukuttan DP. Strategies to manage patients with dental anxiety and dental phobia: literature review. Clin Cosmet Investig Dent. 2016 Mar 10;8:35-50. doi: 10.2147/CCIDE.S63626. eCollection 2016. PMID 27022303
- [Background] Al-Harasi S, Ashley PF, Moles DR, Parekh S, Walters V. Hypnosis for children undergoing dental treatment. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007154. doi: 10.1002/14651858.CD007154.pub2. PMID 20687082
- [Background] Armfield JM, Heaton LJ. Management of fear and anxiety in the dental clinic: a review. Aust Dent J. 2013 Dec;58(4):390-407; quiz 531. doi: 10.1111/adj.12118. PMID 24320894
- [Background] Nigam AG, Marwah N, Goenka P, Chaudhry A. Correlation of general anxiety and dental anxiety in children aged 3 to 5 years: A clinical survey. J Int Oral Health. 2013 Dec;5(6):18-24. Epub 2013 Dec 26. PMID 24453440
- [Background] Najafpour E, Asl-Aminabadi N, Nuroloyuni S, Jamali Z, Shirazi S. Can galvanic skin conductance be used as an objective indicator of children's anxiety in the dental setting? J Clin Exp Dent. 2017 Mar 1;9(3):e377-e383. doi: 10.4317/jced.53419. eCollection 2017 Mar. PMID 28298978
- [Background] Jones LM, Buchanan H. Assessing children's dental anxiety in New Zealand. N Z Dent J. 2010 Dec;106(4):132-6. PMID 21197816
- [Background] Han HR. Measuring anxiety in children: a methodological review of the literature. Asian Nurs Res (Korean Soc Nurs Sci). 2009 Jun;3(2):49-62. doi: 10.1016/S1976-1317(09)60016-5. PMID 25030332
- [Background] Litt MD. A model of pain and anxiety associated with acute stressors: distress in dental procedures. Behav Res Ther. 1996 May-Jun;34(5-6):459-76. doi: 10.1016/0005-7967(96)00015-0. PMID 8687368
- [Background] Wood C, Bioy A. Hypnosis and pain in children. J Pain Symptom Manage. 2008 Apr;35(4):437-46. doi: 10.1016/j.jpainsymman.2007.05.009. Epub 2008 Feb 4. PMID 18243640
- [Background] Jain AA, Yeluri R, Munshi AK. Measurement and assessment of pain in children--a review. J Clin Pediatr Dent. 2012 Winter;37(2):125-36. doi: 10.17796/jcpd.37.2.k84341490806t770. PMID 23534317
- [Background] Kolosovas-Machuca ES, Martinez-Jimenez MA, Ramirez-GarciaLuna JL, Gonzalez FJ, Pozos-Guillen AJ, Campos-Lara NP, Pierdant-Perez M. Pain Measurement through Temperature Changes in Children Undergoing Dental Extractions. Pain Res Manag. 2016;2016:4372617. doi: 10.1155/2016/4372617. Epub 2016 Apr 26. PMID 27445611
- [Background] Seinfeld S, Bergstrom I, Pomes A, Arroyo-Palacios J, Vico F, Slater M, Sanchez-Vives MV. Influence of Music on Anxiety Induced by Fear of Heights in Virtual Reality. Front Psychol. 2016 Jan 5;6:1969. doi: 10.3389/fpsyg.2015.01969. eCollection 2015. PMID 26779081
- [Background] Ramirez-Carrasco A, Butron-Tellez Giron C, Sanchez-Armass O, Pierdant-Perez M. Effectiveness of Hypnosis in Combination with Conventional Techniques of Behavior Management in Anxiety/Pain Reduction during Dental Anesthetic Infiltration. Pain Res Manag. 2017;2017:1434015. doi: 10.1155/2017/1434015. Epub 2017 Apr 11. PMID 28490941
- [Background] Bai J, Hsu L, Tang Y, van Dijk M. Validation of the COMFORT Behavior scale and the FLACC scale for pain assessment in Chinese children after cardiac surgery. Pain Manag Nurs. 2012 Mar;13(1):18-26. doi: 10.1016/j.pmn.2010.07.002. Epub 2011 Feb 24. PMID 22341137
- [Background] Crellin DJ, Harrison D, Santamaria N, Babl FE. Systematic review of the Face, Legs, Activity, Cry and Consolability scale for assessing pain in infants and children: is it reliable, valid, and feasible for use? Pain. 2015 Nov;156(11):2132-2151. doi: 10.1097/j.pain.0000000000000305. PMID 26207651
- [Background] Raslan N, Masri R. A randomized clinical trial to compare pain levels during three types of oral anesthetic injections and the effect of Dentalvibe(R) on injection pain in children. Int J Paediatr Dent. 2018 Jan;28(1):102-110. doi: 10.1111/ipd.12313. Epub 2017 Jun 24. PMID 28646527
- [Background] Johansson M, Kokinsky E. The COMFORT behavioural scale and the modified FLACC scale in paediatric intensive care. Nurs Crit Care. 2009 May-Jun;14(3):122-30. doi: 10.1111/j.1478-5153.2009.00323.x. PMID 19366409
- [Background] Elkins GR, Barabasz AF, Council JR, Spiegel D. Advancing Research and Practice: The Revised APA Division 30 Definition of Hypnosis. Am J Clin Hypn. 2015 Apr;57(4):378-85. doi: 10.1080/00029157.2015.1011465. PMID 25928776
- [Background] Gold JI, Kant AJ, Belmont KA, Butler LD. Practitioner review: clinical applications of pediatric hypnosis. J Child Psychol Psychiatry. 2007 Aug;48(8):744-54. doi: 10.1111/j.1469-7610.2007.01759.x. PMID 17683446
- [Background] Birnie KA, Noel M, Parker JA, Chambers CT, Uman LS, Kisely SR, McGrath PJ. Systematic review and meta-analysis of distraction and hypnosis for needle-related pain and distress in children and adolescents. J Pediatr Psychol. 2014 Sep;39(8):783-808. doi: 10.1093/jpepsy/jsu029. Epub 2014 Jun 2. PMID 24891439
- [Background] Milling LS, Costantino CA. Clinical hypnosis with children: first steps toward empirical support. Int J Clin Exp Hypn. 2000 Apr;48(2):113-37. doi: 10.1080/00207140008410044. PMID 10769980
- [Background] Oberoi J, Panda A, Garg I. Effect of Hypnosis During Administration of Local Anesthesia in Six- to 16-year-old Children. Pediatr Dent. 2016 Mar-Apr;38(2):112-5. PMID 27097858
- [Derived] Giron CB, Ramirez-Carrasco A, Cappello OS, Pozos-Guillen A, Pierdant-Perez M. The efficacy of hypnosis compared with the tell/show/do technique for the reduction of anxiety/pain in children undergoing pulpotomies: a randomized controlled trial. J Clin Pediatr Dent. 2024 Jan;48(1):69-77. doi: 10.22514/jocpd.2024.009. Epub 2024 Jan 3. PMID 38239158